CLINICAL TRIAL: NCT02077296
Title: The Predictive Value of Cytokines on Response to Preoperative Chemoradiotherapy in Patients With Rectal Cancer
Acronym: CYTORECT
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Lotte Jacobs, MD, MD, St. Antonius Hospital
Other Study IDs: NL46983.100.13/R13.044
Record Dates: First submitted 2014-02-26; First posted 2014-03-04 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Cancer
Keywords: cytokines; predictive value; preoperative chemoradiotherapy; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An extra ethylene diamine tetra acetic acid blood tube of 4 ml will be withdrawn from the patient during a regular venapuncture or after administration of an intravenous needle specifically before, during and just after preoperative CRT, 1 day before and 2 days after surgery and 6 weeks after surgery. Blood samples for determination of cytokines are directly processed.
  As standard medical treatment surgery will be performed and biopsies of resection specimen will be collected by the department of pathology, frozen, and further examined. For this study 4 extra biopsies will be taken from resection tissue for cytokine measurements. Two from tumour tissue and 2 from normal mucosa of each patient. These biopsies will be snap-frozen in liquid nitrogen. Subsequently, the frozen biopsies will be grinded with a mortar and pestle, which were cooled in liquid nitrogen, and resuspended in 100 μl ice-cold PBS containing 10 μl/ml of a cocktail of protease inhibitors.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preoperative chemoradiotherapy: The group consists of patients aged ≥18 with a pathohistological diagnosis of locally advanced rectal adenocarcinoma (<15 cm from the anal verge). They are found eligible for preoperative chemoradiotherapy (chemotherapy: oral capecitabine / radiotherapy: 45-50 Gy in total; fractions of 1.8-2 Gy) and surgery (stage 2 or 3 rectal cancer).

SUMMARY:
Rationale and background: Predictive factors are needed to discriminate chemoradiotherapy responders from non-responders and to individualize the treatment regime. Various cytokines play a role in processes affecting tumour growth and metastasis. Furthermore, cytokines might influence treatment response. Various cytokines are abnormally expressed in colorectal cancer patients, are associated with colorectal cancer or determine response to chemoradiotherapy. Therefore the investigators want to investigate whether levels of circulating cytokines could predict response to preoperative chemoradiotherapy in patients with rectal cancer.

Hypothesis: The investigators hypothesis is that the varying levels of circulating cytokines in the blood of rectal cancer patients may predict the response to preoperative chemoradiotherapy.

Study design: This study is an explorative clinical pilot study in which the investigators will collect 4 ml of blood from a selection of rectal cancer patients during a regular venipuncture before, during and after preoperative chemoradiotherapy and before and after surgery. Cytokines will be measured in blood plasma and in tumour and healthy tissue from the resection specimen using multiplex immunoassays. Plasma cytokine measurements will be linked to pathological response to identify which cytokines and corresponding levels can predict response to preoperative chemoradiotherapy for patients with locally advanced rectal cancer. Furthermore, blood plasma cytokine measurements before and after surgery will be compared to evaluate the effect of tumour resection on the immune response. In addition, preoperative blood plasma cytokine levels will be compared with cytokine levels in normal and tumour tissue to test whether circulating cytokine levels are representative for tissue cytokine levels.

Study population: Thirty patients (≥18 years) with locally advanced rectal adenocarcinoma eligible for preoperative chemoradiotherapy (oral capecitabine and 45-50 gray (Gy) in total; fractions of 1.8-2 Gy) and surgery.

Country of recruitment: The Netherlands

ELIGIBILITY:
Inclusion Criteria:

* Pathohistological diagnosis of locally advanced rectal adenocarcinoma (<15 cm from the anal verge)
* Eligible for preoperative chemoradiotherapy (chemotherapy: oral capecitabine / radiotherapy: 45-50 Gy in total; fractions of 1.8-2 Gy) and surgery (stage 2 or 3 rectal cancer)
* Planned to undergo a venipuncture for a regular blood collection during preoperative chemoradiotherapy, before, and after surgery
* Written informed consent
* Age ≥18

Exclusion Criteria:

* Age <18
* Serious adverse events during preoperative chemoradiotherapy
* Use of corticosteroids and/or immunosuppressive drugs during or 1 month prior to the study
* Other malignancies in medical history
* Previous pelvic radiotherapy and/or chemotherapy
* Confirmed bacterial or viral infection during the study or 3 months prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer diagnosed in St. Antonius Hospital Nieuwegein and Utrecht, 18 years or older, selected for preoperative chemoradiotherapy (chemotherapy: oral capecitabine; radiotherapy: 45-50 Gy in total; fractions of 1.8-2 Gy) and surgery. Rectal carcinoma is defined as <15 cm from the anal verge. They are already routinely planned to undergo a regular venipuncture for blood collection and intravenous needle before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Plasma and tissue cytokine levels | 20 weeks
  Patients will be followed for the duration of preoperative chemoradiotherapy until 6 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maartje Los, MD, PhD, Principal Investigator — St. Antonius Hospital; Niels Van Lelyveld, MD, PhD, Principal Investigator — St. Antonius Hospital; G.T. Rijkers, MD, PhD, Prof, Principal Investigator — St. Antonius Hospital; Lotte Jacobs, MD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lin CC, Liu CY, Chen MJ, Wang TE, Chu CH, Wang HY, Shih SC, Hsu ML, Hsu TC, Chen YJ. Profiles of circulating endothelial cells and serum cytokines during adjuvant chemoradiation in rectal cancer patients. Clin Transl Oncol. 2013 Oct;15(10):855-60. doi: 10.1007/s12094-013-1004-6. Epub 2013 Feb 12. PMID 23401019
- [Background] Tsavaris N, Voutsas IF, Kosmas C, Gritzapis AD, Baxevanis CN. Combined treatment with bevacizumab and standard chemotherapy restores abnormal immune parameters in advanced colorectal cancer patients. Invest New Drugs. 2012 Feb;30(1):395-402. doi: 10.1007/s10637-010-9533-0. Epub 2010 Sep 7. PMID 20820907
- [Background] Xynos ID, Karadima ML, Voutsas IF, Amptoulach S, Skopelitis E, Kosmas C, Gritzapis AD, Tsavaris N. Chemotherapy +/- cetuximab modulates peripheral immune responses in metastatic colorectal cancer. Oncology. 2013;84(5):273-83. doi: 10.1159/000343282. Epub 2013 Feb 22. PMID 23445638
- [Background] Trikha M, Corringham R, Klein B, Rossi JF. Targeted anti-interleukin-6 monoclonal antibody therapy for cancer: a review of the rationale and clinical evidence. Clin Cancer Res. 2003 Oct 15;9(13):4653-65. PMID 14581334
- [Background] Kinoshita T, Ito H, Miki C. Serum interleukin-6 level reflects the tumor proliferative activity in patients with colorectal carcinoma. Cancer. 1999 Jun 15;85(12):2526-31. doi: 10.1002/(sici)1097-0142(19990615)85:123.0.co;2-3. PMID 10375098
- [Background] Debucquoy A, Haustermans K, Daemen A, Aydin S, Libbrecht L, Gevaert O, De Moor B, Tejpar S, McBride WH, Penninckx F, Scalliet P, Stroh C, Vlassak S, Sempoux C, Machiels JP. Molecular response to cetuximab and efficacy of preoperative cetuximab-based chemoradiation in rectal cancer. J Clin Oncol. 2009 Jun 10;27(17):2751-7. doi: 10.1200/JCO.2008.18.5033. Epub 2009 Mar 30. PMID 19332731